CLINICAL TRIAL: NCT05153239
Title: A Randomized, Multicenter, Open-label, Phase III Study of Lurbinectedin Single-Agent or Lurbinectedin in Combination With Irinotecan Versus Investigator's Choice (Topotecan or Irinotecan) in Relapsed Small Cell Lung Cancer Patients (LAGOON Trial)
Brief Title: Clinical Trial of Lurbinectedin as Single-agent or in Combination With Irinotecan Versus Topotecan or Irinotecan in Patients With Relapsed Small-cell Lung Cancer (LAGOON)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PM1183-C-008-21
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Relapsed Small Cell Lung Cancer
Keywords: Relapsed Small Cell Lung Cancer; PharmaMar; Lurbinectedin; Irinotecan; Topotecan
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Irinotecan; PM 01183; Topotecan

STUDY DESIGN:
Intervention Model Description: Multicenter, open-label, randomized, controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lurbinectedin (Experimental): Patients will consecutively receive lurbinectedin on Day 1 q3wk (every three weeks = one treatment cycle)
  Interventions: Drug: Lurbinectedin
- Lurbinectedin plus Irinotecan (Experimental): Patients will consecutively receive the following q3wk (every three weeks = one treatment cycle):
  * Irinotecan (Day 1 and Day 8)
  * Lurbinectedin (Day 1)
  Interventions: Drug: Irinotecan; Drug: Lurbinectedin
- Control arm (Active Comparator): Best Investigator's choice prior to randomization between:
  * Irinotecan on Day 1 q3wk
  * Topotecan on Days 1-5 q3wk
  Interventions: Drug: Irinotecan; Drug: Topotecan

INTERVENTIONS:
Drug: Irinotecan — Irinotecan 75 mg/m² intravenously Days 1 & 8 q3wk
  Arms: Lurbinectedin plus Irinotecan
Drug: Lurbinectedin — Lurbinectedin 3.2 mg/m² will be administered intravenously on Day 1 q3wk
  Other Names: PM01183
  Arms: Lurbinectedin
Drug: Irinotecan — For patients aged <70 years: irinotecan 350 mg/m² intravenously Day 1 q3wk For patients aged ≥70 years: irinotecan 300 mg/m² intravenously Day 1 q3wk
  Arms: Control arm
Drug: Topotecan — Topotecan 2.3 mg/m² oral or 1.5 mg/m² intravenously Days 1-5 q3wk
  Arms: Control arm
Drug: Lurbinectedin — Lurbinectedin 2.0 mg/m² will be administered intravenously on Day 1 q3wk
  Other Names: PM01183
  Arms: Lurbinectedin plus Irinotecan

SUMMARY:
Multicenter, open-label, randomized, controlled phase III clinical trial to evaluate and compare the activity and safety of two experimental arms consisting of lurbinectedin as single agent (Group A) or the combination of lurbinectedin with irinotecan (Group B) versus Investigator's Choice (topotecan or irinotecan) as control arm (Group C), in Small-cell Lung Cancer (SCLC) patients who failed one prior platinum-containing line.

DETAILED DESCRIPTION:
Approximately 705 Adult SCLC patients with Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 2 who have failed one prior platinum-containing line with CTFI ≥ 30 days and controlled asymptomatic and pretreated Central Nervous System metastases will be enrolled and assigned to each treatment arm.

Central randomization will be implemented; patients will be assigned to each treatment arm at a 1:1:1 ratio.

An Independent Data Monitoring Committee (IDMC) will oversee the conduct of the study. The IDMC should have access to unblinded efficacy and safety data throughout the trial to enable timely and informed judgments about risks and benefits.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent of the patient obtained before any study-specific procedure
2. Age≥18 years
3. Histologically or cytologically confirmed diagnosis of SCLC.
4. One prior line of platinum-containing chemotherapy with/without anti-PD-1 or anti-PD-L1 (Note: at least 70% of patients included in the study have to be pretreated with anti-PD-1 or anti-PD-L1)
5. Chemotherapy-free interval (CTFI, time from the last dose of first-line platinum-containing chemotherapy to the occurrence of progressive disease) ≥ 30 days (independent of the immunotherapy maintenance, if applicable)
6. Patients with history of Central Nervous System (CNS) metastases can participate provided they are pretreated and radiologically stable (i.e., without evidence of progression) for at least 4 weeks by repeated imaging (note: repeated imaging should be performed during study screening), asymptomatic, and without requirement of steroid treatment for at least 7 days before the first dose of study treatment
7. Eastern Cooperative Oncology Group (ECOG) PS ≤ 2
8. Adequate hematological, renal, metabolic and hepatic function:

   1. Hemoglobin ≥ 9.0 g/dL [patients may have received prior red blood cell (RBC) transfusion, if clinically indicated]; absolute neutrophil count (ANC) ≥ 2.0 x 10^9/L, and platelet count ≥ 100 x 10^9/L.
   2. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3.0 x upper limit of normal (ULN).
   3. Total bilirubin ≤ 1.5 x ULN or direct bilirubin ≤ ULN.
   4. Albumin ≥ 3.0 g/dL.
   5. Calculated creatinine clearance (CrCL) ≥ 30 mL/min (using Cockcroft and Gault's formula).
9. At least three weeks since last prior antineoplastic treatment and recovery to grade ≤ 1 from any adverse event (AE) related to previous anticancer treatment (excluding sensory neuropathy, immune-related hypothyroidism, anemia, asthenia and alopecia, all grade ≤ 2) according to the National Cancer InstituteCommon Terminology Criteria for Adverse Events (NCICTCAE) v.5.
10. Prior radiotherapy (RT): At least two weeks since completion of prophylactic cranial irradiation (PCI), and to any other site not previously specified.
11. Evidence of non-childbearing status for women of childbearing potential (WOCBP). WOCBP must agree to use a highly effective contraceptive measure up to seven months after treatment discontinuation. Fertile male patients with WOCBP partners should use condoms during treatment and for four months following the last investigational medicinal product (IMP) dose.

Exclusion Criteria:

1. Platinum-naïve patients or patients pretreated with more than one prior chemotherapy regimen (including patients re-challenged with same initial regimen).
2. Prior treatment with lurbinectedin, trabectedin, PM14, or topoisomerase I inhibitors (irinotecan, topotecan, etc.).
3. Active or untreated CNS metastases and/or carcinomatous meningitis.
4. Patients with limited-stage disease who are candidates for local or regional therapy, including PCI, thoracic RT or both, must have been offered that option and completed treatment or refused it prior to randomization.
5. Concomitant diseases/conditions:

   1. History or presence of unstable angina, myocardial infarction, congestive heart failure, or clinically significant valvular heart disease within last year.
   2. Symptomatic arrhythmia or any uncontrolled arrhythmia requiring ongoing treatment.
   3. Ongoing chronic alcohol consumption or cirrhosis with Child-Pugh score B or C.
   4. Known Gilbert's disease.
   5. Active uncontrolled infection. Serious non-healing wound, ulcer or bone fracture. Presence of external drainages.
   6. Ongoing, treatment-requiring, non-neoplastic chronic liver disease of any origin. For Hepatitis B, this includes positive tests for both Hepatitis B surface antigen (HBsAg) and quantitative Hepatitis B polymerase chain reaction (PCR). For Hepatitis C, this includes positive tests for both Hepatitis C antibody and quantitative Hepatitis C PCR. Subjects taking hepatitis related antiviral therapy within six months prior to the first dose of study drugs will also be excluded.
   7. Intermittent or continuous oxygen requirement within two weeks prior to randomization. Patients with confirmed or suspected diagnosis of diffuse interstitial lung disease or pulmonary fibrosis.
   8. Patients with a second invasive malignancy treated with chemotherapy and/or RT. Patients with a previous malignancy that was completely resected with curative intention three or more years prior to randomization, except treated in situ carcinoma of the cervix, basal or squamous cell skin carcinoma, and in situ transitional cell bladder carcinoma and who has been continuously in remission since then will be permitted.
   9. Limitation of the patient's ability to comply with the treatment or to follow the protocol.
   10. Documented or suspected invasive fungal infections requiring systemic treatment within 12 weeks of randomization.
   11. Known human immunodeficiency virus (HIV) infection.
   12. Any past or present chronic inflammatory colon and/or liver disease, past intestinal obstruction, pseudo or subocclusion or paralysis.
   13. Evident symptomatic pleural or cardiac effusion rapidly increasing and/or necessitating prompt local treatment within seven days.
   14. Any other major illness that, in the Investigator's judgment, will substantially increase the risk associated with the patient's participation in this study (e.g.; COVID-19 disease).
6. RT in more than 35% of the bone marrow.
7. History of previous bone marrow and/or stem cell transplantation and allogenic transplant.
8. Patient has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of inactivated vaccines is allowed.
9. Impending need for RT (e.g., painful bone metastasis and/or risk of spinal cord compression).
10. History of allergy or hypersensitivity to any of the study drugs or any of their excipients.
11. Women who are pregnant or breast feeding and fertile patients (men and women) who are not able to use a highly effective method of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 705 (Estimated)
Dates: Start 2022-07-22 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From the date of randomization to the date of death or last contact, up to 39 months
  Overall survival (OS) will be calculated from the date of randomization to the date of death or last contact (in this case, survival will be censored on that date).

SECONDARY OUTCOMES:
Progression-free survival by IRC (Independent Review Committee) | From the date of randomization to the date of progressive disease, death or last tumor assessment or further anticancer treatment, up to 39 months
  Progression-free survival (PFS) will be calculated from the date of randomization to the date of documented progression per RECIST v.1.1 (Progressive disease is declared when there is an increase in sum of target disease ≥ 20%) or death (regardless of the cause of death). If the patient receives further antitumor therapy, withdraws from the study, or is lost to follow-up before progressive disease (PD), PFS will be censored at the date of last evaluable tumor assessment before the date of subsequent antitumor therapy.
Progression-free survival by IA (Investigator Assessment) | From the date of randomization to the date of progressive disease, death or last tumor assessment or further anticancer treatment, up to 39 months
  Progression-free survival (PFS) will be calculated from the date of randomization to the date of documented progression per RECIST v.1.1 (Progressive disease is declared when there is an increase in sum of target disease ≥ 20%) or death (regardless of the cause of death). If the patient receives further antitumor therapy, withdraws from the study, or is lost to follow-up before progressive disease (PD), PFS will be censored at the date of last evaluable tumor assessment before the date of subsequent antitumor therapy.
Overall response rate by IRC | From the date of randomization to the date of death or last contact, up to 39 months
  Overall response rate (ORR) will be the percentage of patients with complete or partial response as the best response obtained in any evaluation according to RECIST v.1.1. Progressive disease is declared when there is an increase in sum of target disease ≥ 20%, stable disease when the change is > -30% and ≤ 20%, partial response when there is a decrease in sum of target disease ≥ 30%, and complete response when all lesions have disappeared or all lesions have disappeared and all nodal disease is < 10 mm each.
Overall response rate by IA | From the date of randomization to the date of death or last contact, up to 39 months
  Overall response rate (ORR) will be the percentage of patients with complete or partial response as the best response obtained in any evaluation according to RECIST v.1.1. Progressive disease is declared when there is an increase in sum of target disease ≥ 20%, stable disease when the change is > -30% and ≤ 20%, partial response when there is a decrease in sum of target disease ≥ 30%, and complete response when all lesions have disappeared or all lesions have disappeared and all nodal disease is < 10 mm each.
Overall survival rate at 12 months | At 12 months
  Overall survival rate at 12 months is defined as the percentage of people who are still alive at 12 months after randomization.
Overall survival rate at 24 months | At 24 months
  Overall survival rate at 24 months is defined as the percentage of people who are still alive at 24 months after randomization.
Progression-free survival rate at 6 months by IRC | At 6 months
  Progression-free survival rate at 6 months is defined as the percentage of people who remain free from progression at 6 months after randomization
Progression-free survival rate at 6 months by IA | At 6 months
  Progression-free survival rate at 6 months is defined as the percentage of people who remain free from progression at 6 months after randomization
Progression-free survival rate at 12 months by IRC | At 12 months
  Progression-free survival rate at 12 months is defined as the percentage of people who remain free from progression at 12 months after randomization
Progression-free survival rate at 12 months by IA | At 12 months
  Progression-free survival rate at 12 months is defined as the percentage of people who remain free from progression at 12 months after randomization
Duration of response by IRC | From the date of first documentation of complete or partial response to the date of documented progression disease, death or last contact, up to 39 months
  Duration of response (DoR) will be calculated from the date of first documentation of response per RECIST v.1.1 (complete or partial response, whichever occurs first) to the date of documented PD or death. Progressive disease is declared when there is an increase in sum of target disease ≥ 20%, stable disease when the change is > -30% and ≤ 20%, partial response when there is a decrease in sum of target disease ≥ 30%, and complete response when all lesions have disappeared or all lesions have disappeared and all nodal disease is < 10 mm each.
Duration of response by IA | From the date of first documentation of complete or partial response to the date of documented progression disease, death or last contact, up to 39 months
  Duration of response (DoR) will be calculated from the date of first documentation of response per RECIST v.1.1 (complete or partial response, whichever occurs first) to the date of documented PD or death. Progressive disease is declared when there is an increase in sum of target disease ≥ 20%, stable disease when the change is > -30% and ≤ 20%, partial response when there is a decrease in sum of target disease ≥ 30%, and complete response when all lesions have disappeared or all lesions have disappeared and all nodal disease is < 10 mm each.
Patient-reported outcomes | At baseline and every six weeks (± one week) until end of treatment, up to 39 months
  To measure the quality of life of patients, the Lung Cancer Symptom Scale (LCSS) questionnaire will be analyzed.

CONTACTS AND LOCATIONS:
Locations (210):
- United States (15):
  - Ironwood Cancer & Research Centers, Chandler, Arizona
  - Genesis Cancer and Blood, Hot Springs, Arkansas
  - Florida Cancer Specialists - South, Fort Myers, Florida
  - Florida Cancer Specialists - North, St. Petersburg, Florida
  - Florida Cancer Specialists - Panhandle, Tallahassee, Florida
  - Florida Cancer Specialists - East, West Palm Beach, Florida
  - Duly Health and Care, Joliet, Illinois
  - Norton Cancer Institue, Downtown, Louisville, Kentucky
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Oncology Hematology West, PC (Grand Island), Grand Island, Nebraska
  - Oncology Hematology West, PC dba Nebraska Cancer Specialists, Omaha, Nebraska
  - FirstHealth Outpatient Cancer Center, Pinehurst, North Carolina
  - Utah Cancer Specialists, Salt Lake City, Utah
  - MultiCare Regional Cancer Center - Tacoma, Tacoma, Washington
  - Froedtert Hospital/Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (8):
  - The Chris Obrien Lifehouse, Camperdown, New South Wales
  - BRICC - Ballarat Health Services, Ballarat Central, Victoria
  - Box Hill Hospital Eastern Health Clinical School, Box Hill, Victoria
  - Northern Beaches Hospital, Frenchs Forest
  - Gosford Hospital GH - Central Coast Cancer Centre, Gosford
  - Austin Hospital- Medical Oncology Unit, Heidelberg
  - St John of God Murdoch Hospital, Murdoch
  - Cancer Care Wollongong, Wollongong
- Austria (2):
  - University Hospital Salzburg, Salzburg
  - Medizinische Universitaet Wien, Vienna
- Belgium (8):
  - Antwerp University Hospital, Edegem, Antwerp
  - Algemeen Ziekenhuis AZ Klina - Borstkliniek, Brasschaat
  - Grand Hopital de Charleroi GHdC - Hopital Saint Joseph, Charleroi
  - Centre Hospitalier Chretien CHC - MontLegia, Liège
  - CHR de la Citadelle, Liège
  - CHU Liege, Liège
  - Az Sint Maarten Mechelen, Mechelen
  - Centre Hospitalier Universitaire (CHU) Ambroise Pare, Mons
- Brazil (8):
  - Oncocentro-Centro de Oncologia do Parana, Curitiba, Paraná
  - UPCO - Hospital de Clinicas de Porto Alegre, Santa Cecília, Porto Alegre
  - Nucleo de Oncologia da Bahia - NOB, Ondina, Salvador
  - Fundacao Pio XII - Hospital de Cancer de Barretos - Hospital de Amor, Barretos
  - ONCOSITE - Centro de Pesquisa Clinica em Oncologia Ltda, Ijuí
  - Irmandade daSanta Casa de Misericordia de Porto Alegre, Porto Alegre
  - Hospital Sao Lucas da PUCRS, Porto Alegre
  - Instituto Nacional de Cancer - Ministrio da Sade, Rio de Janeiro
- Bulgaria (4):
  - Multiprofile Hospital for Active Treatment - Uni Hospital OOD Department of Medical Oncology, Panagyurishte
  - Complex Oncology Center - Plovdiv EOOD, First Department of Medical Oncology and Oncological Diseases in Gastroenterology, Plovdiv
  - Specialized hospital for active treatment of oncological diseases, Sofia
  - Multiprofile Hospital for Active Treatment Serdika EOOD Second Department of Medical Oncology, Sofia
- Canada (6):
  - Hamilton Health Sciences -Juravinski Cancer Centre, Hamilton, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Hôpital de la Cité-de-la- Santé, Laval, Quebec
  - CISSS de la Montérégie-Centre - Hôpital Charles LeMoyne, Longueuil, Quebec
  - McGill University Health Centre (MUHC), Montreal
  - University Health Network - Princess Margaret Hospital, Toronto
- Chile (7):
  - Clinical Research Chile SpA, Valdivia, Los Ríos Region
  - James Lind Centro de Investigación del Cáncer, Temuco, Región de la Araucanía
  - Centro de Estudios Clínicos SAGA, Santiago
  - Clinica Alemana de Santiago, Santiago
  - Clínica Santa María, Santiago
  - Fundación Arturo López Pérez, Santiago
  - Hospital Clinico Universidad de Chile, Santiago
- Denmark (4):
  - Aalborg University Hospital, Aalborg
  - Sjællands Universitetshospital, Næstved
  - Sønderborg Sygehus, Sønderborg
  - Vejle Hospital, Vejle
- France (13):
  - Hopital Jean Minjoz, Besançon
  - AssAP-HP - Hopital Ambroise-Pare, Boulogne-Billancourt
  - Hopital Morvan CHU de Brest, Brest
  - Centre François Baclesse, Caen
  - CHU de Caen - Hopital Cote de Nacre, Caen
  - Centre Hospitalier Intercommunal de Creteil (CHIC), Créteil
  - Centre Hospitalier Universitaire CHU De Limoges, Limoges
  - CHU de Nantes, Nantes
  - Bichat-Claude Bernard Hospital, Paris
  - CHU Reims - Hpital Maison Blanche, Reims
  - Hopital Civil / Nouvel Hopital Civil, Strasbourg
  - Hospital Foch, Suresnes
  - Gustave Roussy, Villejuif
- Georgia (6):
  - High Technology Hospital Medcenter, Batumi
  - Todua Clinic, Tbilisi
  - New Hospitals, Tbilisi
  - Institute Of Clinical Oncology, Tbilisi
  - JSC Evex Hospitals "Caraps Medline", Tbilisi
  - LTD Cancer Research Centre, Tbilisi
- Germany (17):
  - LungenClinic Grosshansdorf, Großhansdorf, Schleswig-Holstein
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Evangelische Lungenklinik Berlin, Berlin
  - Klinikum Bremen Ost, Bremen
  - Helios St. Johannes Klinikum, Duisburg
  - Klinikum Esslingen GmbH, Esslingen am Neckar
  - Universittsklinikum Freiburg, Freiburg im Breisgau
  - Asklepios Fachklinik München-Gauting, Gauting
  - Krankenhaus Martha-Maria Halle gGmbH, Halle
  - Universitaetsklinikum Halle Saale, Halle
  - Thoraxclinic Heidelberg GmbH, Heidelberg
  - Vincentius-Diakonissen-Kliniken gAG Karlsruhe, Karlsruhe
  - Klinikum Kassel - Medizinische Klinik IV, Kassel
  - Klinik Loewenstein gGmbH, Löwenstein
  - Universitaetsmedizin Mannheim, Mannheim
  - Staedtisches Klinikum München - Bogenhausen, München
  - Sana Klinikum Offenbach, Offenbach
- Hungary (5):
  - Debreceni Egyetem - Klinikai Kozpont, Debrecen
  - Veszprem Megyei Tudogyogyintezet Farkasgyepu, Farkasgyepű
  - Bacs-Kiskun County Hospital, Kecskemét
  - Hetenyi G Korhaz, Onkologiai Kozpont, Szolnok
  - Pulmonology Hospital Torokbalint, Törökbálint
- Israel (5):
  - Rambam Health Care Campu, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - The Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (19):
  - A.O. SS. Antonio e Biagio e Cesare Arrigo di Alessandria, Alessandria
  - Azienda Ospedaliero Universitaria delle Marche, Ancona
  - IRCCS Centro di Riferimento Oncologico, Aviano
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna Policlinico S. Orsola Malpighi Oncologia medica, Bologna
  - Azienda Ospedaliera Univ. Policlinico G Rodolico San Marco, Catania
  - A.O. Santa Croce e Carle, Ospedale Carle, Cuneo
  - AOU Careggi, Florence
  - ASL 3 Genovese Oncologia Medica Villa Scassi, Genova
  - IRCCS Istituto Clinico Humanitas - Cancer Center, Milan
  - Universita degli Studi della Campania Luigi Vanvitelli, Napoli
  - Ospedale Maggiore di Novara, Novara
  - Azienda Ospedaliero-Universitaria San Luigi Gonzaga, Orbassano
  - Oncologia Medica II Istituto Oncologico Veneto IRCCS, Padua
  - Azienda USL di Piacenza, Piacenza
  - Irccs-Crob, Rionero in Vulture
  - Fondazione Policlinico Universitario Campus Bio-Medico, Roma
  - IFO Regina Elena, Roma
  - ASST Valtellina e Alto Lario Ospedale di Sondrio, Sondrio
  - ASST Sette Laghi, Varese
- Japan (14):
  - Hirosaki University Hospital, Hirosaki, Aomori
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Ohara HealthCare Foundation Kurashiki Central Hospital, Kurashiki, Okayama-ken
  - Osaka Habikino Medical Center, Habikino, Osaka
  - Kansai Medical University Hospital, Hirakata-shi, Osaka
  - Izumi City General Hospital, Izumi, Osaka
  - Kanagawa Cancer Center, Izumi, Osaka
  - Kishiwada City Hospital, Kishiwada, Osaka
  - Tokyo Metropolitan Cancer and Infectious Diseases Center Komagome Hospital, Bunkyō-Ku, Tokyo
  - The Cancer Institute Hospital Of JFCR, Koto-Ku, Tokyo
  - Center Hospital of the National Center for Global Health and Medicine, Shinjuku-Ku, Tokyo
- Poland (7):
  - II Klinika Chorob Pluc i Gruzlicy, Bialystok
  - Szpitale Pomorskie Sp. z o.o., Oddzial Onkologii K, Gdynia
  - Wojewódzkie Wielospecjalistyczne Centrum Onkologii, Lodz
  - Specjalistyczna Praktyka Lekarska Slawomir Mandziuka, Lublin
  - Szpital Specjalistyczny w Prabutach Sp. z o.o, Prabuty
  - Mrukmed. Lekarz Beata Madej-Mruk i Partner. Sp.p, Rzeszów
  - Specjalistyczny Szpital Onkologiczny NU-MED sp. Z, Tomaszów Mazowiecki
- Romania (6):
  - Sc Oncopremium Team Srl, Baia Mare
  - Medisprof srl, Cluj-Napoca
  - Oncolab SRL, Craiova
  - Centrul de Oncologie Sfantu Nectarie, Craiova
  - Ovidius Clinical Hospital, Ovidiu
  - Oncocenter Oncologie clinica S.R.L, Timișoara
- South Korea (9):
  - Chungbuk National University Hospital, Cheongju-si
  - CHA Bundang Medical Center, CHA University, Gyeonggi-do
  - The Catholic University of Korea, St.Vincents Hospital, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Kangbuk Samsung Hospital, Seoul
  - Asan Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Seoul Metropolitan Government-Seoul National University Boramae Medical Center, Seoul
- Spain (24):
  - Institut Català d Oncologia (ICO) - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Institut Catala d'Oncologia (ICO) - Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Complejo Hospitalario Materno-Insular de Gran Canaria, Las Palmas de Gran Canaria, Gran Canaria
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Complexo Hospitalario Universitario De Vigo (CHUVI) - Hospital Xeral, Vigo, Pontevedra
  - Hospital Teresa Herrera C.H.U.A., A Coruña
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Universitario La Paz, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Clínica Universidad de Navarra, Madrid
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Fundación Jimenez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Regional Universitario Málaga Hospital Civil, Málaga
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitari i Politècnic La Fe, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Hospital Clínico Universitario Lozano Bleza, Zaragoza
- Switzerland (7):
  - University Hospital Basel, Basel
  - Istituto Oncologico della Svizzera Italiana, Bellinzona
  - Spital Thurgau - Kantonspital Frauenfeld, Frauenfeld
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital Baselland, Liestal
  - Spital Thurgau - Kantonsspital Muensterlingen, Münsterlingen
  - HFR Freiburg Kantonsspital, Villars-sur-Glâne
- Taiwan (4):
  - Buddhist Dalin Tzu Chi Hospital, Dalin, Chiayi
  - Changhua Christian Hospital, Chang-hua
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - National Taiwan University Cancer Center, Taipei
- Turkey (Türkiye) (5):
  - Medicalpark Seyhan Hospital, Seyhan, Adana
  - Liv Hospital Ankara, Çankaya, Ankara
  - Bagcilar Medipol Mega University Hospital, Bağcılar, Istanbul
  - Goztepe Prof. Dr. Suleyman Yalcin City Hospital, Kadıköy, Istanbul
  - Kocaeli University Hospital, İzmit, Kocaeli
- United Kingdom (7):
  - Belfast Health and Social Care Trust, Belfast
  - The Princess Alexandra Hospital, Harlow
  - Guys and St Thomas NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - Clatterbridge Hospital, Metropolitan Borough of Wirral
  - Nottingham University Hospitals NHS Trust, Nottingham
  - The Royal Wolverhampton NHS Trust, Wolverhampton